CLINICAL TRIAL: NCT01340768
Title: An Open-Label, Randomized Naturalistic Study to Evaluate the Incidence of Hypoglycemia Comparing Sitagliptin With Sulfonylurea Treatment in Patients With Type 2 Diabetes During Ramadan Fasting
Brief Title: Study to Compare Sitagliptin Versus Sulfonylurea Treatment During Ramadan Fasting in Patients With Type 2 Diabetes (MK-0431-262)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-262; CTRI/2011/06/001838 (Registry Identifier: CTRI)
Record Dates: First submitted 2011-03-24; First posted 2011-04-25 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glucose metabolism disorders Metabolic diseases Peptidase inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Sulfonylurea Compounds; glimepiride; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100mg taken orally once daily with or without metformin
  Interventions: Drug: Sitagliptin; Drug: Metformin
- Sulfonylurea Therapy (Active Comparator): Usual sulfonylurea therapy with or without metformin
  Interventions: Drug: Sulfonylurea; Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin — One 100 mg tablet taken orally once daily
  Other Names: Sitagliptin phosphate, MK-0431, JANUVIA®
  Arms: Sitagliptin
Drug: Sulfonylurea — Participant continued pre-study sulfonylurea therapy (dose as prescribed by the physician). Pre-study sulfonylurea therapy consisted of either glibenclamide, glimepiride or gliclazide.
  Other Names: Amaryl (glimepiride)
  Arms: Sulfonylurea Therapy
Drug: Metformin — Participants receiving metformin at enrollment, continued pre-study doses of metformin. If necessary, the physician could either discontinue or adjust the dose of metformin during Ramadan.
  Other Names: Glucophage

SUMMARY:
This is a study comparing the incidence of hypoglycemia while using sitagliptin treatment versus sulfonylurea (SU) treatment in participants with type 2 diabetes mellitus (T2DM) who regularly take an SU drug, and choose to fast during the month of Ramadan. The primary hypothesis is that during the 30 days of Ramadan fasting, treatment with sitagliptin (with or without metformin) compared to SU treatment (with or without metformin) results in a lower incidence of hypoglycemia in participants with T2DM.

DETAILED DESCRIPTION:
This study and NCT01131182 (MK-0431-263) have the same design but are conducted under separate protocols, in different countries, according to local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Muslim, with type 2 diabetes mellitus
* Intends to fast during the month of Ramadan
* Hemoglobin A1c (HbA1c) ≤10% at screening
* On a stable dose of a SU drug (glibenclamide, glimepiride, or gliclazide), for at least three months, with or without metformin therapy at a stable dose

Exclusion Criteria:

* Type 1 diabetes mellitus
* Pregnant or breast feeding or with gestational diabetes
* Hypersensitivity or contraindication to dipeptidyl peptidase-4 (DPP-4) treatment
* Serum creatinine ≥1.5 mg/dL (males), ≥1.4 mg/dL (females)
* History of severe hypoglycemia (defined as a hypoglycemic event requiring the assistance of another individual, and/or resulting in a emergency department admission, physician office visit and/or hospitalization)
* Any use of insulin (prior to or during Ramadan)
* Use of any class of oral antidiabetic therapy other than an SU or metformin
* Current participation in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2010-06-22 (Actual); Primary Completion 2011-09-21 (Actual); Study Completion 2011-09-21 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Lee SWH, Chen WS, Sellappans R, Md Sharif SB, Metzendorf MI, Lai NM. Interventions for people with type 2 diabetes mellitus fasting during Ramadan. Cochrane Database Syst Rev. 2023 Jul 12;7(7):CD013178. doi: 10.1002/14651858.CD013178.pub2. PMID 37435938
- [Derived] Aravind SR, Ismail SB, Balamurugan R, Gupta JB, Wadhwa T, Loh SM, Suryawanshi S, Davies MJ, Girman CJ, Katzeff HL, Radican L, Engel SS, Wolthers T. Hypoglycemia in patients with type 2 diabetes from India and Malaysia treated with sitagliptin or a sulfonylurea during Ramadan: a randomized, pragmatic study. Curr Med Res Opin. 2012 Aug;28(8):1289-96. doi: 10.1185/03007995.2012.707119. Epub 2012 Jul 6. PMID 22738801

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin: Sitagliptin 100mg taken orally once daily, with or without metformin
- Sulfonylurea Therapy: Usual sulfonylurea therapy and dose for each participant, with or without metformin
Period: Overall Study
Arm/Group | Sitagliptin | Sulfonylurea Therapy
Started | 436 | 434
Completed | 419 | 429
Not Completed | 17 | 5
Not completed — Lost to Follow-up | 10 | 4
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin: Sitagliptin 100mg taken orally once daily with or without metformin. All participants as treated population defined as all randomized participants who received at least one dose of study drug.
- Sulfonylurea Therapy: Usual sulfonylurea therapy and dose for each participant, with or without metformin. All participants as treated population defined as all randomized participants who received at least one dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Sulfonylurea Therapy | Total
Number analyzed (Participants) | 421 | 427 | 848
Age, Continuous [Mean (Full Range); unit: years] | 51.4 [26 to 80] | 50.7 [23 to 78] | 51.0 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 233 | 446
  Male | 208 | 194 | 402

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Symptomatic Hypoglycemic Event
Description: Symptomatic hypoglycemic events were based on the participants own self-reported symptoms (for example, but not limited to the following: faintness, headache, confusion, anxiety, sweating, tremor, palpitations, nausea, pallor, dizziness, hunger, sudden behavioral change).
Time Frame: Up to 30 days (Day 1 through last day of Ramadan)
Population: All participants as treated population defined as all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Sitagliptin | Sulfonylurea Therapy
Number analyzed (Participants) | 421 | 427
percentage of participants | 3.8 | 7.3
Statistical Analysis 1: Comparison: Sitagliptin vs Sulfonylurea Therapy; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel — P-value for association between treatment groups and proportions controlling for prior therapy (monotherapy or combination therapy); Risk Ratio (RR) = 0.52, 95% CI 2-sided [0.29 to 0.94]

2. Secondary Outcome: Percentage of Participants With at Least One Symptomatic or Asymptomatic Hypoglycemic Event
Description: Symptomatic hypoglycemic events were based on the participants own self-reported symptoms (for example but not limited to the following: faintness, headache, confusion, anxiety, sweating, tremor, palpitations, nausea, pallor, dizziness, hunger, sudden behavioral change). Asymptomatic hypoglycemic events were based on self-monitored finger-stick blood glucose level.
Time Frame: Up to 30 days (Day 1 through last day of Ramadan)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Sitagliptin | Sulfonylurea Therapy
Number analyzed (Participants) | 421 | 427
percentage of participants | 4.8 | 9.6
Statistical Analysis 1: Comparison: Sitagliptin vs Sulfonylurea Therapy; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.29 to 0.83]

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Sulfonylurea Therapy
Serious Adverse Events (participants affected / at risk) | 1/421 | 0/427
Other Adverse Events (participants affected / at risk) | 16/421 | 33/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=421) | Sulfonylurea Therapy (N=427)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=421) | Sulfonylurea Therapy (N=427)
Hypoglycemia (Metabolism and nutrition disorders) | 16 (19) | 33 (63) — Hypoglycemia includes both symptomatic hypoglycemia and asymptomatic hypoglycemia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall not publish any article or paper nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations, relating or referring to the following: (a) the study or any results, data or insight there from; (b) the services performed; or (c) any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of the sponsor.